CLINICAL TRIAL: NCT06970288
Title: Effectiveness of Introducing Ultra-High B-Value Diffusion-Weighted Imaging as a Modified Abbreviated Protocol for Breast Cancer Detection
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD45/2025
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the added value of non-contrast abbreviated MRI protocol featuring ultra-high B value Diffusion Weighted Imaging to detect, characterize suspicious breast lesions and avoid using contrast.

ELIGIBILITY:
Inclusion Criteria:

* • Women with suspicious breast mass (BIRADS 4a)

  * High risk women (Positive family history)
  * Women with suspicious axillary lymph nodes by Ultrasound
  * Women with dense breasts coming for MRI imaging.

Exclusion Criteria:

* • Contraindications to MRI

  * Pacemaker, cochlear implant, claustrophobia, ocular implants
  * Contraindications to contrast administration:
  * Elevated kidney functions
  * Women who haven't undergone reliable Mammogram & Ultrasound
  * Women with prior treatment or intervention (e.g. biopsy)
  * Patients' refusal.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women in childbearing age who have a suspicious breast lump
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the capability of detecting suspicious breast lesions using non-contrast enhanced MRI protocol featuring ultra-high B-value | 20 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt